CLINICAL TRIAL: NCT04718467
Title: A Single-center, Randomized, Double-Blinded, Placebo-Controlled, Phase Ⅱb Clinical Trial of Recombinant COVID-19 Vaccine (Sf9 Cells), in the Subjects From Healthy Aged 18 to 85 Years Old
Brief Title: Phase IIb Clinical Trial of Recombinant Novel Coronavirus Pneumonia (COVID-19) Vaccine (Sf9 Cells)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to cancel this trial.
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT107
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: Safety; Immunogenicity; COVID-19 Vaccine; Recombinant vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- adults group (aged 18-59 years) & vaccine (Experimental): three doses of 40μg Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21, 42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cells)
- adults group (aged 18-59 years) & placebo (Placebo Comparator): three doses of placebo at the schedule of day 0, 21, 42.
  Interventions: Biological: Placebo
- elderly adults group (aged 60-85 years) & vaccine (Experimental): three doses of 40μg Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21, 42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cells)
- elderly adults group (aged 60-85 years) & placebo (Placebo Comparator): three doses of placebo at the schedule of day 0, 21, 42.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant COVID-19 vaccine (Sf9 cells) — Three doses of Recombinant COVID-19 vaccine (Sf9 cells) (40μg) at the schedule of day 0, 21, 42.
  Arms: adults group (aged 18-59 years) & vaccine; elderly adults group (aged 60-85 years) & vaccine
Biological: Placebo — Three doses of Placebo (1.0ml) at the schedule of day 0, 21, 42.
  Arms: adults group (aged 18-59 years) & placebo; elderly adults group (aged 60-85 years) & placebo

SUMMARY:
This is a phase Ⅱb, single-center, randomized, double-blind, placebo-controlled study, to evaluate the immunogenicity and safety of the recombinant COVID-19 vaccine (Sf9 cells) in the subjects from healthy adults and elderly adults aged 18 years and above (aged 18-59 and 60-85 years) with immunization procedures 0, 21, 42 days and doses 40μg.

DETAILED DESCRIPTION:
This is a phase Ⅱb, single-center, randomized, double-blind, placebo-controlled study, to evaluate the immunogenicity and safety of the recombinant COVID-19 vaccine (Sf9 cells) in the subjects from healthy adults and elderly adults aged 18 years and above (aged 18-59 and 60-85 years) . The phase Ⅱb clinical trials designed two research group, including adults group (aged 18-59 years) and elderly adults group (aged 60-85 years). Each group including 2000 participants. Vaccination or placebo group will be randomly assigned to receive in a 3:1 ratio, 4000 in total.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85 years old
* Able to understand the content of informed consent and willing to sign the informed consent.
* Able and willing to complete all the secluded study process during the whole study follow-up period (about 14 months).
* Axillary temperature ≤37.0℃

Exclusion Criteria:

* Positive serum immunoglobulin M (IgM) and immunoglobulin G (IgG) to the SARS-CoV-2.
* SARS-CoV-2 nucleic acid testing positive.
* History of SARS-CoV-2 infection or vaccination
* A Known History of HIV infection
* Family history of seizure, epilepsy, brain or mental disease.
* Participant that has an allergic history to any ingredient of vaccines.
* Woman who is pregnant, breast-feeding or positive in pregnancy test on day of enrollment, or is planning to be pregnant during the next 14 months.
* Any acute fever disease or infections.
* Have a medical history of SARS.
* Have serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension and not well-controlled.
* Major chronic illness, such as asthma, diabetes, or thyroid disease, and not well-controlled.
* Malignant tumor, activity or have been treated tumor and no clear have cured, or during the study period is likely to relapse.
* Hereditary angioneurotic edema or acquired angioneurotic edema.
* Urticaria in last one year.
* Asplenia or functional asplenia.
* Platelet disorder or other bleeding disorder may cause injection contraindication.
* Faint at the sight of blood or needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylactics treatment, cytotoxic treatment in last 6 months.
* Prior administration of blood products in last 4 months.
* Prior administration of other research medicines in last 1 month.
* Prior administration of attenuated vaccine in last 1 month.
* Prior administration of subunit vaccine or inactivated vaccine in last 14 days.
* Nearly 7 days, all sorts of acute onset of disease or chronic diseases, such as receiving anti-tuberculosis treatment, history of asthma.
* According to the investigator's judgment, due to various medical, psychological, social or other conditions, it is contrary to the trial protocol or affects the subjects to sign informed consent.

Exclusion criteria for subsequent doses:

* Appear systemic allergic reaction, severe allergic reactions.
* Appear difficult to tolerate more than grade 3 adverse reactions.
* New discovery or a new happened after the first vaccination does not conform to the first dose of the inclusion criteria or conform to the first dose of exclusion criteria, determine whether or not to continue to participate in the study by the investigators.
* Investigators think of other reasons.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse reaction (AR) | 0 to 7 days after each dose
  The incidence of adverse reaction (AR)
The incidence of Adverse Events of Special Interest (AESI) | from day 0 to day 60 after last dose
  The incidence of Adverse Events of Special Interest (AESI)

SECONDARY OUTCOMES:
The incidence of adverse events (AE) | from day 0 to day 30 after last dose
  The incidence of adverse events (AE)
The incidence of grade 3 adverse events (AE) | from day 0 to day 30 after last dose
  The incidence of grade 3 adverse events (AE)
The incidence of severe adverse events (SAE) | Month 12 after the whole process of vaccination
  The incidence of severe adverse events (SAE)
Geometric mean (GMT) of specific antibody | day 30, day 60, month 6, month 12 after last dose
  Geometric mean (GMT) of specific antibody against Severe Acute Respiratory Syndrome Coronavirus 2 (SARSCoV-2) Spike protein Receptor-binding domain(S-RBD) protein (ELISA) in immunogenicity subgroup.
Geometric mean (GMT) of anti-SARS-CoV-2-specific neutralizing antibodies | day 30, day 60, month 6, month 12 after last dose
  Geometric mean (GMT) of anti-SARS-CoV-2-specific neutralizing antibodies (euvirus and pseudovirus-neutralizing assays)
The positive conversion rate of S-RBD protein-specific antibody | day 30, day 60, month 6, month 12 after last dose
  The positive conversion rate of S-RBD protein-specific antibody (ELISA) against SARS-CoV-2
Geometric mean fold increase (GMI) of S-RBD protein-specific antibody | day 30, day 60, month 6, month 12 after last dose
  Geometric mean fold increase (GMI) of S-RBD protein-specific antibody (ELISA) against SARS-CoV-2
The positive conversion rate of anti-SARS-CoV-2 specific neutralizing antibody | day 30, day 60, month 6, month 12 after last dose
  The positive conversion rate of anti-SARS-CoV-2 specific neutralizing antibody (euvirus and pseudovirus neutralization test)
Geometric mean fold increase (GMI) of anti-SARS-CoV-2 specific neutralizing antibodies | day 30, day 60, month 6, month 12 after last dose
  Geometric mean fold increase (GMI) of anti-SARS-CoV-2 specific neutralizing antibodies (eucivirus and pseudovirus neutralization assays)

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Doctor, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China